CLINICAL TRIAL: NCT04965337
Title: A Phase I Randomized, Double-Blind, Placebo-Controlled, Dose Escalation, Single Center Bridging Study to Evaluate Safety, Tolerability and Pharmacokinetics of ASC42 in Chinese Healthy Subjects
Brief Title: Study to Evaluate Safety, Tolerability and Pharmacokinetics of ASC42 in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ASC42-102
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: Healthy Subjects; ASC42; FXR agonist

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ASC42 Dose A (Experimental): ASC42 tablet Dose A, once daily
  Interventions: Drug: ASC42
- Placebo Dose A (Placebo Comparator): Placebo Comparator: Single dose of matched placebo to ASC42 tablet Dose A, once daily
  Interventions: Drug: Placebo
- ASC42 Dose B (Experimental): ASC42 tablet Dose B, once daily
  Interventions: Drug: ASC42
- Placebo Dose B (Placebo Comparator): Placebo Comparator: Single dose of matched placebo to ASC42 tablet Dose A, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASC42 — ASC42 tablet administered orally
  Arms: ASC42 Dose A; ASC42 Dose B
Drug: Placebo — Matching placebo administered orally
  Arms: Placebo Dose A; Placebo Dose B

SUMMARY:
This is a Phase I Randomized, Double-Blind, Placebo-Controlled, Dose Escalation, Single Center Bridging Study to Evaluate Safety, Tolerability and Pharmacokinetics of ASC42 in Chinese Healthy Subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male and female volunteers aged 18-55 years.
* 19kg/m2 ≤ BMI <24kg/m2.

Key Exclusion Criteria:

* A positive HBsAg, HCV Ab and/or HIV Ab.
* Pancreatic injury or pancreatitis.
* History of organ transplantation, including bone marrow transplantation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-11 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
AUC of ASC42 | Up to 4 days
  Evaluate the Area under the plasma concentration versus time curve.
Cmax of ASC42 | Up to 4 days
  Evaluate the Peak Plasma Concentration.

SECONDARY OUTCOMES:
t1/2 of ASC42 | Up to 4 days
  Evaluate the Terminal-Phase Half-Life.
CL/F of ASC42 | Up to 4 days
  Evaluate the Apparent Systemic Clearance.
Vd/F of ASC42 | Up to 4 days
  Evaluate the Apparent Volume of Distribution.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 7 days
  Occurrence of Serious Adverse Event (SAE), Adverse Event (AE) resulting in treatment discontinuation and/or dose reductions, and AE of special interest, from baseline up to 7 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Boai Rehabilitation Hospital, Changsha, Hunan, China